CLINICAL TRIAL: NCT02506972
Title: Effect of Varying Amounts of β-glucan and Sucrose in Oatmeal on Glycemic Response
Brief Title: Effect of Serving Size and Addition of Sugar on the Glycemic Response Elicited by Oatmeal
Acronym: Panther
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glycemic Index Laboratories, Inc (Industry)
Collaborators: PepsiCo Global R&D (Industry); Applied Statistics and Consulting (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GIL-1404
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus
Keywords: Blood glucose; Humans; Postprandial; Sugar; Carbohydrate; Oat beta-glucan
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- 30g oats (Other): Classic Quick Quaker Oats
  Interventions: Other: Classic Quaker Quick Oats
- 30g oats plus 9g sugar (Other): Classic Quick Quaker Oats
  Interventions: Other: Classic Quaker Quick Oats
- 40g oats (Other): Classic Quick Quaker Oats
  Interventions: Other: Classic Quaker Quick Oats
- 60g oats (Other): Classic Quick Quaker Oats
  Interventions: Other: Classic Quaker Quick Oats
- 22g cream of rice cereal (Other): Cream of Rice Cereal, B&G Foods, Inc.
  Interventions: Other: Cream of Rice Cereal
- 29g cream of rice cereal (Other): Cream of Rice Cereal, B&G Foods, Inc.
  Interventions: Other: Cream of Rice Cereal
- 33g cream of rice cereal (Other): Cream of Rice Cereal, B&G Foods, Inc.
  Interventions: Other: Cream of Rice Cereal
- 44g cream of rice cereal (Other): Cream of Rice Cereal, B&G Foods, Inc.
  Interventions: Other: Cream of Rice Cereal

INTERVENTIONS:
Other: Classic Quaker Quick Oats — Various doses of oats without or with sugar
  Arms: 30g oats; 30g oats plus 9g sugar; 40g oats; 60g oats
Other: Cream of Rice Cereal — Various doses of cereal without sugar
  Arms: 22g cream of rice cereal; 29g cream of rice cereal; 33g cream of rice cereal; 44g cream of rice cereal

SUMMARY:
The purpose of this study was to determine the impact of serving size and the addition of sugar on the glycemic response elicited by oatmeal compared to that elicited by cream of rice cereal.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) 20.0 - 34.9 kg/m²

Exclusion Criteria:

* known to have diabetes
* use of medications considered by the principal investigator to influence glycemic responses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Incremental area under the blood glucose response curve | For 2 hours after consuming each test meal

SECONDARY OUTCOMES:
Peak rise of blood glucose | During 2 hour period after consuming each test meal
  The highest concentration of blood glucose achieved after eating minus the fasting blood glucose.
Time to peak | During 2 hour period after consuming each test meal
  The time at which the peak rise of blood glucose occured.
Mean rate of decline in blood glucose | During 2 hour period after consuming each test meal
  The rate of change in blood glucose between consecutive time points (Tx and T(x+1)) was calculated as: Rx = (Gx G(x+1))/(Tx-T(x+1)), where G(x+1) and Gx were the glucose concentrations at times T(x+1) and Tx, respectively. The mean rate of decline in blood glucose (Mean RD) was calculated as the weighted average of all the Rx values from the time of the peak glucose concentration to 120 min, with the weight based on the length of the time interval.
Maximum rate of decline in blood glucose | During 2 hour period after consuming each test meal
  The rate of change in blood glucose between consecutive time points (Tx and T(x+1)) was calculated as: Rx = (Gx G(x+1))/(Tx-T(x+1)), where G(x+1) and Gx were the glucose concentrations at times T(x+1) and Tx, respectively. . The maximum rate in blood glucose decline (Max RD) was calculated as the maximum of all the Rx values from the time of the peak glucose concentration to 120 min.
Time to baseline | During 2 hour period after consuming each test meal
  The time for blood glucose to return to baseline was linearly interpolated between the first blood glucose concentration below fasting and the previous value; if blood glucose did not reach baseline, Bt was taken to be 120min.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Inc., Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wolever TMS, van Klinken BJ, Spruill SE, Jenkins AL, Chu Y, Harkness L. Effect of serving size and addition of sugar on the glycemic response elicited by oatmeal: A randomized, cross-over study. Clin Nutr ESPEN. 2016 Dec;16:48-54. doi: 10.1016/j.clnesp.2016.07.003. Epub 2016 Sep 1. PMID 28531455